CLINICAL TRIAL: NCT05813977
Title: Is it Possible to Decrease Droplet Generation During Percutaneous Dilatational Tracheotomy?
Brief Title: Amount of Droplet Formed During Percutaneous Dilatational Tracheostomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Diskapi Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Eda Macit Aydın, Principal Investigator, specialist, intensivisit, Ankara Diskapi Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Droplet
Record Dates: First submitted 2023-03-09; First posted 2023-04-14 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Ventilatory Failure
Keywords: Percutaneous Dilatational Tracheotomy; Flow controlled ventilation; droplet
MeSH Terms: conditions — Hypoventilation

STUDY DESIGN:
Intervention Model Description: Group 1: Tritube (FCV) Group 2: Conventional endotracheal tube
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1: Tritube (FCV) used during tracheostomy (Experimental): The patient is intubated with Tritube® after the removal of the conventional endotracheal tube (ETT) and Tritube® was advanced until proximal to the carina. Before starting the PDT, measurements with ATP bioluminescence-based method (3M Clean-trace®) were made by taking sample from a sterile PVC (poly vinyl chloride) surface (10 cm2) which is held 50 cm over the operation site. After PDT with Griggs method (Portex), the measurements were repeated by taking sample from surface.
  Interventions: Device: tritube
- Group 2: Conventional endotracheal tube used during tracheostomy (No Intervention): In the patient who was intubated with a conventional endotracheal tube (ETT), the tube was withdrawal to the vocal cords. Before starting the PDT, measurements with ATP bioluminescence-based method (3M Clean-trace®) were made by taking sample from a sterile PVC surface (10 cm2) which is held 50 cm over the operation site. After PDT with Griggs method (Portex), the measurements were repeated by taking sample from surface.

INTERVENTIONS:
Device: tritube — The patient is intubated with Tritube® after the removal of the conventional endotracheal tube (ETT) and Tritube® was advanced until proximal to the carina. Before starting the PDT, measurements with ATP bioluminescence-based method (3M Clean-trace®) were made by taking sample from a sterile PVC surface (10 cm2) which is held 50 cm over the operation site. After PDT with Griggs method (Portex), the measurements were repeated by taking sample from surface.
  Arms: Group 1: Tritube (FCV) used during tracheostomy

SUMMARY:
During the percutaneous dilatational tracheostomy (PDT), large amount of droplets and aerosols are spread to the environment especially with the effect of ventilation during the dilatation phase. In such cases, it is recommended to take precautions such as masks and goggles or shields to protect practitioners from infection, however it has also been reported that droplets and aerosols can spread to the environment and can go far.

Flow controlled ventilation (FCV) with the use of Tritube® and Evone® could reduce droplet spread during PDT and provide a safer environment while operating on patients with infected airways.

DETAILED DESCRIPTION:
During the percutaneous dilatational tracheostomy, large amount of droplets and aerosols are spread to the environment especially with the effect of ventilation during the dilatation phase. In such cases, it is recommended to take precautions such as masks and goggles or shields to protect practitioners from infection, however it has also been reported that droplets and aerosols can spread to the environment and can go far.

Flow controlled ventilation (FCV) with the use of Tritube® and Evone® could reduce droplet spread during PDT and provide a safer environment while operating on patients with infected airways.

SPSS 21.0 (Statistical Package for the Social Sciences) (Version 22.0, SPSS, Inc, Chicago, USA) program will be used for statistical analysis. After applying the Shapiro-wilk test for normality, the student's t test will be used if the distribution is not normal. Fisher's exact test or chi-square test will be used for categorical variables. Results p<0.05 will be considered significant.

The investigators compared the amount of droplets scattered in the environment with PDT performed with FCV and conventional mechanical ventilation methods, with the ATP (adenosine triphosphate) bioluminescence method.

ELIGIBILITY:
Inclusion Criteria:

* percutaneous tracheostomy procedure

Exclusion Criteria:

* whose written consent cannot be obtained
* who undergo surgical tracheostomy for any reason
* patients with active infection in the area of the procedure

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2023-04-11 (Actual); Primary Completion 2023-09-14 (Actual); Study Completion 2023-09-14 (Actual)

PRIMARY OUTCOMES:
the outcome measures (droplet account) are assessing a change | 1th min before sterilization and 1th min after tracheostomy cannula insertion
  The investigators hypothesized that droplet account will decrease while tritube using

SECONDARY OUTCOMES:
complication rates | 24 hour after tracheostomy procedure
  the complications such as endotracheal tube (ET) cuff puncture, Difficult insertion of tracheostomy tube, Accidental extubation, Bleeding vs. during percutaneous tracheostomy

CONTACTS AND LOCATIONS:
Overall Officials: Eda MACİT AYDIN, Principal Investigator — Ankara Diskapi Training and Research Hospital
Locations (1):
- Diskapi Training and Resource Hospital, Ankara, Ankara, Turkey (Türkiye)